CLINICAL TRIAL: NCT06581731
Title: Comparison of the Safety and Effectiveness of Remifentanil with a Combination of Remimazolam and Dexmedetomidine for Awake Fibreoptic Nasotracheal Intubation
Brief Title: Comparison of Remifentanil with a Combination of Remimazolam and Dexmedetomidine for Awake Tracheal Intubation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY20240514-01
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-05

CONDITIONS: Difficult or Failed Intubation; Sedative Adverse Reaction
Keywords: AFOI; Dexmedetomidine; Rimazazolam; Remifentanil
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group remimazolam-remifentanil (Experimental): Administer 5 mg of remimazolam intravenously, followed by a continuous infusion at a rate of 0.5 mg/kg/h to maintain anesthesia.
  Interventions: Drug: remimazolam combined with remifentanil; Drug: dexmedetomidine combined with remifentanil
- group dexmedetomidine-remifentanil (Experimental): Administer 1 μg/kg of dexmedetomidine as an intravenous bolus over 10 minutes, followed by a continuous infusion at 0.5 μg/kg/h to maintain anesthesia.
  Interventions: Drug: remimazolam combined with remifentanil; Drug: dexmedetomidine combined with remifentanil

INTERVENTIONS:
Drug: remimazolam combined with remifentanil — Patients in this group will receive a bolus of remimazolam 5 mg intravenously, and then a dose of 0.1 μg/kg/min remifentanil and 0.5 mg/kg/h remimazolam via separate syringe pumps.
  Other Names: remimazolam-remifentanil
Drug: dexmedetomidine combined with remifentanil — Patients in this group will receive a loading dose of dexmedetomidine 1 μg/kg over 10 minutes intravenously, and then a dose of 0.1 μg/kg/min remifentanil and 0.5 μg/kg/h dexmedetomidine via separate syringe pumps.
  Other Names: dexmedetomidine-remifentanil

SUMMARY:
Awake fiberoptic intubation (AFOI) requires airway surface anesthesia to inhibit pharyngeal reflex, glottis closure reflex, and cough reflex. Additionally, the use of sedative drugs can enhance patient comfort and tolerance, reduce anxiety, and eliminate harmful effects on systemic hemodynamics.The objective of this study is to compare the safety and efficacy of remifentanil alone versus a combination of dexmedetomidine and remifentanil for sedation during conscious tracheal intubation.

DETAILED DESCRIPTION:
Awake fiberoptic intubation (AFOI) is regarded as the gold standard for managing anticipated difficult airways due to its high success rate and low risk. However, awake intubation can induce significant stress responses in patients, including increased heart rate, severe blood pressure fluctuations, and intense coughing. Therefore, during awake intubation, airway local anesthesia techniques are necessary to suppress the gag reflex, glottic closure reflex, and cough reflex, enabling the patient to tolerate the stress responses associated with intubation. In addition to local anesthesia, sedatives are typically required to enhance patient comfort and tolerance, reduce anxiety, and minimize adverse effects on systemic hemodynamics. However, excessive sedation can lead to complications such as airway collapse, hypoxemia, and respiratory depression, while insufficient sedation may result in severe coughing and discomfort. The ideal sedative state preserves spontaneous breathing, maintains low sensitivity to nausea and vomiting, and allows for awakening if necessary. Safety and comfort are the primary considerations in selecting sedative medications; therefore, sedative and analgesic drugs used in AFOI should be short-acting, easily titratable, and minimally suppressive of spontaneous respiration.The most commonly used sedatives include benzodiazepines, propofol, remifentanil, and dexmedetomidine. During AFOI, a combination of the two drugs can be used to meet the requirements of sedation and analgesia. Remifentanil has a fast onset, fast elimination, and does not rely on liver and kidney function. It is the first ultra short acting opioid drug in clinical practice, and its termination of action is not significantly related to infusion time and dose. It provides sufficient analgesia and good anesthesia controllability for patients with difficult airway during conscious intubation. Rimazolen is an ester metabolite derivative of the benzodiazepine drug midazolam, which has been successfully used for the induction and maintenance of programmed sedation and general anesthesia due to its fast onset, short duration of sedative effect, and short recovery time, with a half-life of 5-10 minutes. In addition, remifentanil has no effect on heart rate, electrocardiogram, blood pressure, and respiratory rate. Rimazolen accumulates rarely after long-term infusion and does not affect liver and kidney function, making it safe for patients with liver or kidney dysfunction. In addition, remifentanil sedation can be reversed by flumazenil, and it may be a useful medication in clinical situations that require maintenance of spontaneous ventilation. Research reports that the combination of benzodiazepines and opioids may be an ideal drug for AFOI. Dexmedetomidine is a highly selective α 2-adrenergic agonist that produces dose-dependent sedative and anti anxiety effects, with a certain degree of analgesic effect. It can preserve airway reflex, dilate tracheal smooth muscle, and inhibit cough response without causing respiratory depression. However, it may cause bradycardia, heart block, and hypotension, and has a slow onset when used alone. Dexmedetomidine has a rapid onset of action and a terminal half-life of 2 hours. It is metabolized in the liver and its metabolites are eliminated through urine. Therefore, the dosage should be reduced appropriately in patients with renal or liver dysfunction. Dexmedetomidine combined with opioid drugs is also commonly used for AFOI.

There is currently no consensus on the safest and most effective sedative drugs for conscious tracheal intubation, and using a single drug often fails to meet all the requirements of Awake Fiberoptic Intubation (AFOI). The ideal sedative should provide effective conscious sedation while maintaining autonomous ventilation, ensuring smooth intubation conditions, and stabilizing hemodynamics. Therefore, the objective of this study is to compare the safety and efficacy of remifentanil alone versus a combination of dexmedetomidine and remifentanil for sedation during conscious tracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing general anesthesia who require awake nasal tracheal intubation.
2. Age 18-65 years old
3. ASA classifications of I-III
4. BMI<30kg/m2

Exclusion Criteria:

1. Patients allergic to propofol, midazolam, dexmedetomidine, remifentanil.
2. Second- or third-degree atrioventricular block, rate <50 beats/min, systolic blood pressure <90 mmHg
3. Acute exacerbation of respiratory diseases such as asthma, bronchitis, and chronic obstructive pulmonary disease (COPD)
4. Patients with acute arrhythmias and severe heart disease (congenital, valvular diseases)
5. Patients with severe liver or kidney dysfunction requiring replacement therapy
6. Patients with severe mental disorders requiring medication for symptom control and experiencing communication barriers
7. Patients with moderate to severe anemia, coagulation disorders, and hematologic diseases
8. Patients with basal skull fractures, facial fractures, significantly deviated nasal septum, or nasal cavity diseases causing severe nasal congestion
9. patients on long-term opioids or sedative medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
intubation scores | preoperative
  Perform a four-level scoring based on vocal cord movement (open, movement, closed), cough intensity (none, mild, moderate, severe), and limb movement (none, mild, moderate, severe).
intubation comfort scores | preoperative
  patient tolerance was assessed by intubation comfort scores (1, no reaction, no change or a single change in the facial expression; 2, slight reaction, grimacing facial expressions; 3, moderate reaction, severe facial grimace but retained ability to follow verbal command and no reflex head movements; 4 severe reaction, severe facial grimace associated with head movements, but patient remains able to obey verbal commands; 5, very severe reaction, severe facial grimace associated with protective head and limb movements hindering the procedure and an inability to obey any verbal command; 6, uncooperative)

SECONDARY OUTCOMES:
hypoxia | intraoperative
  SPO2<90%
occurrence of adverse reactions other than hypoxia | intraoperative
  hypertension, hypotension, tachycardia, bradycardia
clinical outcome immediately following the Awake Fiberoptic Intubation | intraoperative
  1, cooperative; 2, restless with minimal resistance; 3, severe resistance with immediate application of general anesthesia
recall of the Awake Fiberoptic Intubation | after surgery, up to 24h
  1 = none, 2 = partial, and 3 = full
satisfaction score of the Awake Fiberoptic Intubation | after surgery, up to 24h
  1 = excellent, 2 = good, 3 = acceptable, and 4 = poor

CONTACTS AND LOCATIONS:
Overall Officials: Hongwei Shi, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China